CLINICAL TRIAL: NCT00107172
Title: A Randomized Phase III Study of Sublobar Resection Versus Sublobar Resection Plus Brachytherapy in High Risk Patients With Non-Small Cell Lung Cancer (NSCLC), 3cm or Smaller
Brief Title: Surgery With or Without Internal Radiation Therapy in Treating Patients With Stage I Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACOSOG-Z4032; ACOSOG-Z4032; CDR0000422346 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Results first posted 2016-12-23 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative; Brachytherapy

ARMS (2):
- Arm I (Active Comparator): Patients undergo open or thoracoscopic sublobar resection comprising either a wedge resection or anatomical segmentectomy.
  Interventions: Procedure: surgery
- Arm II (Experimental): Patients undergo surgery as in arm I. Patients also undergo intraoperative brachytherapy comprising an iodine I 125 implant at the resection margin.
  Interventions: Procedure: surgery; Radiation: brachytherapy

INTERVENTIONS:
Procedure: surgery
Radiation: brachytherapy
  Arms: Arm II

SUMMARY:
This randomized phase III trial studies surgery and internal radiation therapy to see how well they work compared to surgery alone in treating patients with stage I non-small cell lung cancer. Surgery may be an effective treatment for non-small cell lung cancer. Internal radiation uses radioactive material placed directly into or near a tumor to kill tumor cells. It is not yet known whether surgery and internal radiation therapy are more effective than surgery alone in treating non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To ascertain whether patients treated by sublobar resection (SR) + brachytherhapy (BX) have longer time to local recurrence as compared to the patients treated by SR (local recurrence includes recurrence within the same lobe or hilum [N1 nodes], or progression at the staple line after treatment effects such as scarring have subsided).

SECONDARY OBJECTIVES:

I. To compare procedure specific morbidity and mortality between study arms. II. To compare overall survival and failure-free survival between study arms. III. To assess freedom from regional or distant recurrence. IV. To assess the effect of histological or cytologic positive resection margins on time to local recurrence.

V. To determine the effect of brachytherapy on quality of life (QoL). VI. To determine the effect of brachytherapy on pulmonary function.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo open or thoracoscopic sublobar resection comprising either a wedge resection or anatomical segmentectomy.

ARM II: Patients undergo surgery as in arm I. Patients also undergo intraoperative brachytherapy comprising iodine I 125 implant at the resection margin.

After completion of study treatment, patients are followed at 3, 6, 12, 18, 24, 30, and 36 months and then yearly for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* PART I: PRE-OPERATIVE CRITERIA (PRE-REGISTRATION/RANDOMIZATION)
* Patients must have a suspicious lung nodule for clinical stage I non-small cell lung cancer (NSCLC)
* Patient must have a mass =< 3 cm maximum diameter by computed tomography (CT) size estimate: clinical stage Ia or selected Ib (i.e., with visceral pleural involvement)
* Patient must have a CT scan of the chest with upper abdomen within 60 days prior to date of pre-registration
* Eastern Cooperative Oncology Group (ECOG)/Zubrod performance status 0, 1, or 2
* Patient must meet at least one major criteria or meet a minimum of two minor criteria as described below:

  * Major criteria

    * Forced expiratory volume in 1 second (FEV1) =< 50% predicted
    * Diffusing capacity of the lungs for carbon monoxide (DLCO) =< 50% predicted
  * Minor criteria

    * Age >= 75
    * FEV1 51-60% predicted
    * DLCO 51-60% predicted
    * Pulmonary hypertension (defined as a pulmonary artery systolic pressure greater than 40 mmHg) as estimated by echocardiography or right heart catheterization
    * Poor left ventricular function (defined as an ejection fraction of 40% or less)
    * Resting or exercise partial pressure of oxygen (pO2) =< 55 mm Hg or peripheral capillary oxygen saturation (SpO2) =< 88%
    * Partial pressure of carbon dioxide (pCO2) > 45 mm Hg
    * Modified Medical Research Council (MMRC) Dyspnea Scale >= 3
* Patient must not have had previous intra-thoracic radiation therapy
* Women of child-bearing potential must have negative serum or urine pregnancy test
* No prior invasive malignancy, unless disease-free for >= 5 years prior to pre-registration (exceptions: non-melanoma skin cancer, in-situ cancers)
* PART II: INTRA-OPERATIVE CRITERIA (REGISTRATION)
* Patient must have biopsy-proven NSCLC
* Patient must have all suspicious mediastinal lymph nodes (> 1 cm short-axis dimension on CT scan or positive on positron emission tomography [PET] scan) assessed by one of the following methods to confirm negative involvement with NSCLC (mediastinoscopy, endo-esophageal ultrasound guided needle aspiration, CT-guided, video-assisted thoracoscopic or open lymph node biopsy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2005-07 (Actual); Primary Completion 2013-04-18 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiran C. Fernando, MD, Study Chair — Boston Medical Center
Locations (38):
- United States (37):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - University of California Davis Cancer Center, Sacramento, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Evanston Hospital, Evanston, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Simmons Cooper Cancer Institute, Springfield, Illinois
  - Cancer Institute at St. Joseph Medical Center, Towson, Maryland
  - Boston University Cancer Research Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Valley Hospital - Ridgewood, Ridgewood, New Jersey
  - South Nassau Communities Hospital, Oceanside, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Jameson Memorial Hospital - North Campus, New Castle, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - U.T. Medical Center Cancer Institute, Knoxville, Tennessee
  - Methodist Hospital, Houston, Texas
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Floyd and Delores Jones Cancer Institute at Virginia Mason Medical Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
- London Regional Cancer Program at London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Smith RP, Schuchert M, Komanduri K, Burton S, Heron DE, Luketich JD, d'Amato T, Landreneau R. Dosimetric evaluation of radiation exposure during I-125 vicryl mesh implants: implications for ACOSOG z4032. Ann Surg Oncol. 2007 Dec;14(12):3610-3. doi: 10.1245/s10434-007-9624-0. Epub 2007 Oct 2. PMID 17909906
- [Result] Fernando HC, Landreneau RJ, Mandrekar SJ, Hillman SL, Nichols FC, Meyers B, DiPetrillo TA, Heron DE, Jones DR, Daly BD, Starnes SL, Tan A, Putnam JB. Thirty- and ninety-day outcomes after sublobar resection with and without brachytherapy for non-small cell lung cancer: results from a multicenter phase III study. J Thorac Cardiovasc Surg. 2011 Nov;142(5):1143-51. doi: 10.1016/j.jtcvs.2011.07.051. Epub 2011 Aug 26. PMID 21872277
- [Result] Fernando HC, Landreneau RJ, Mandrekar SJ, Hillman SL, Nichols FC, Meyers B, DiPetrillo TA, Heron D, Jones DR, Daly BD, Starnes SL, Hatter JE, Putnam JB. The impact of adjuvant brachytherapy with sublobar resection on pulmonary function and dyspnea in high-risk patients with operable disease: preliminary results from the American College of Surgeons Oncology Group Z4032 trial. J Thorac Cardiovasc Surg. 2011 Sep;142(3):554-62. doi: 10.1016/j.jtcvs.2010.10.061. Epub 2011 Jul 2. PMID 21724195
- [Result] Fernando HC, Landreneau RJ, Mandrekar SJ, Nichols FC, Hillman SL, Heron DE, Meyers BF, DiPetrillo TA, Jones DR, Starnes SL, Tan AD, Daly BD, Putnam JB Jr. Impact of brachytherapy on local recurrence rates after sublobar resection: results from ACOSOG Z4032 (Alliance), a phase III randomized trial for high-risk operable non-small-cell lung cancer. J Clin Oncol. 2014 Aug 10;32(23):2456-62. doi: 10.1200/JCO.2013.53.4115. Epub 2014 Jun 30. PMID 24982457
- [Result] Fernando HC, Landreneau RJ, Mandrekar SJ, Nichols FC, DiPetrillo TA, Meyers BF, Heron DE, Hillman SL, Jones DR, Starnes SL, Tan AD, Daly BD, Putnam JB; Alliance for Clinical Trials in Oncology. Analysis of longitudinal quality-of-life data in high-risk operable patients with lung cancer: results from the ACOSOG Z4032 (Alliance) multicenter randomized trial. J Thorac Cardiovasc Surg. 2015 Mar;149(3):718-25; discussion 725-6. doi: 10.1016/j.jtcvs.2014.11.003. Epub 2014 Nov 13. PMID 25500100

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two hundred twenty-four (224) participants were accrued between January 2006 and January 2010.
Pre-assignment Details: One participant on SR arm was enrolled from a site with a regulatory violation and 1 participant on SR+BX arm had no surgery. These two participants were excluded from all analyses.
Groups:
- Arm A (SR): Patients undergo open or thoracoscopic sublobar resection (SR) comprising either a wedge resection or anatomical segmentectomy.
- Arm B (SR + BX): Patients undergo sublobar resection plus brachytherapy (SR + BX)
Period: Overall Study
Arm/Group | Arm A (SR) | Arm B (SR + BX)
Started | 114 | 108
Completed | 109 | 103
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 0 | 2
Not completed — Other Reason | 4 | 3

BASELINE CHARACTERISTICS:
Population: All intent-to-treat (ITT) participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (SR) | Arm B (SR + BX) | Total
Number analyzed (Participants) | 114 | 108 | 222
Age, Continuous [Median (Full Range); unit: years] | 70 [49 to 85] | 72 [50 to 87] | 71 [49 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 59 | 124
  Male | 49 | 49 | 98
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 1 | 1
  United States | 114 | 107 | 221
Eastern Cooperative Oncology Group (ECOG)Performance Status [Number; unit: participants]
  0 = Asymptomatic and fully active | 20 | 25 | 45
  1= Symptomatic and fully ambulatory | 66 | 60 | 126
  2= Symptomatic and ambulatory | 28 | 23 | 51
Clinical Nodule Size (cm) [Number; unit: participants]
  <= 2 cm | 73 | 67 | 140
  > 2 cm | 41 | 41 | 82
Tumor Stage [Number; unit: participants] — Tumor staging was defined by tumor location and size. T1=surrounded by lung/visceral pleura, without bronchoscopic evidence of invasion more proximal than the lobar bronchus.
  T2=tumor involves main bronchus, >=2cm distal to the carina; invades the visceral pleura; associated with atelectasis/obstructive pneumonitis that extends to the hilar region but does not involve the entire lung.
  T3=tumor directly invades chest wall, diaphragm, mediastinal pleura, parietal pericardium; tumor in the main bronchus <2cm distal to the carina but without involvement of the carina;
  participants
    T1=Tumor <=3cm | 114 | 104 | 218
    T2=Tumor > 3cm | 0 | 3 | 3
    T3=Tumor of any size | 0 | 1 | 1
Metastatis stage, M0 [Number; unit: participants] — Metastasis stage refers to which organs the cancer has spread. M0 = No distant metastasis
  participants | 114 | 108 | 222
Nodal Stage, N0 [Number; unit: participants] — Nodal stage refers to regional lymph node involvement. N0=No regional lymph node metastasis.
  participants | 114 | 108 | 222
Baseline diffusing capacity of the lung for carbon monoxide (DLCO) [Median (Full Range); unit: Percentage of predicted] | 47 [18 to 97] | 45 [8 to 137] | 46 [8 to 137]
Baseline Forced Expiratory Volume in 1 second (FEV1) [Median (Full Range); unit: Percentage of Predicted] | 48 [22 to 117] | 53 [25 to 110] | 50 [22 to 117]

OUTCOME MEASURES:

1. Primary Outcome: Time to Local Recurrence
Description: Local recurrence included the recurrence within the same lobe or hilum (N1 nodes), or progression at the staple line after treatment effects such as scarring have subsided. Time to local recurrence was censored 1) at the time of a distant recurrence, 2) at the last follow-up time when a patient died within 3 years of randomization without a local recurrence or 3) at 3 years follow-up if the patient remains alive 3 years post-randomization without a local recurrence.
Time Frame: Up to 3 years
Population: All intent-to-treat (ITT) participants.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm A (SR) | Arm B (SR + BX)
Number analyzed (Participants) | 114 | 108
years | NA [NA to NA] — The median and 95% confidence interval to local recurrence has not been attained because of the insufficient number of participants with events. | NA [NA to NA] — The median and 95% confidence interval of time to local recurrence has not been attained because of the insufficient number of participants with events.
Statistical Analysis 1: Comparison: Arm A (SR) vs Arm B (SR + BX); The competing risk analysis accounting for death/regional and distant recurrence as competing events was performed; Test type: Superiority or Other; p = 0.98, Log Rank; Competing risk P-value = 0.91; Cox Proportional Hazard = 1.01, 95% CI 2-sided [0.51 to 1.98]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: Up to 5 years
Population: All intent-to-treat (ITT) participants
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm A (SR) | Arm B (SR + BX)
Number analyzed (Participants) | 114 | 108
years | 5.3 [3.8 to NA] — The upper limit of 95% confidence interval of median survival time has not been attained because of the insufficient number of participants with events. | 4.7 [3.9 to NA] — The upper limit of 95% confidence interval of median survival time has not been attained because of the insufficient number of participants with events.
Statistical Analysis 1: Comparison: Arm A (SR) vs Arm B (SR + BX); Test type: Superiority or Other; p = 0.75, Log Rank; Cox Proportional Hazard = 1.07, 95% CI 2-sided [0.71 to 1.61]

3. Secondary Outcome: Number of Participants Reported Local Recurrence at 3 Years
Description: Local recurrence was defined as the recurrence within the same lobe or hilum (N1 nodes), or at the staple line after treatment effects such as scarring have subsided.
Time Frame: 3 years
Population: All intent-to-treat participants.
Measure: Number; unit: participants
Arm/Group | Arm A (SR) | Arm B (SR + BX)
Number analyzed (Participants) | 114 | 108
participants | 14 | 13

4. Secondary Outcome: Number of Participants Reported Regional Recurrence at 3 Years
Description: Regional recurrence was defined as the recurrence within another lobe or pleura on the same side as the resection, or the ipsilateral mediastinal (N2) nodes.
Time Frame: 3 years
Population: All intent-to-treat participants.
Measure: Number; unit: participants
Arm/Group | Arm A (SR) | Arm B (SR + BX)
Number analyzed (Participants) | 114 | 108
participants | 8 | 9

5. Secondary Outcome: Number of Participants Reported Distant Recurrence at 3 Years
Description: Distant recurrence was defined as the recurrence within contralateral lobe, contralateral mediastinal (N3) nodes or distant> metastatic disease (other organs).
Time Frame: 3 years
Population: All intent-to-treat participants.
Measure: Number; unit: participants
Arm/Group | Arm A (SR) | Arm B (SR + BX)
Number analyzed (Participants) | 114 | 108
participants | 10 | 12

6. Secondary Outcome: Mortality Rates at 30- and 90-day After Sublobar Resection
Time Frame: 90 days
Population: All Intent-to-Treat (ITT) participants
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (SR) | Arm B (SR + BX)
Number analyzed (Participants) | 114 | 108
percentage of participants
  0 - 30 days | 0.9 | 1.9
  0 - 90 days | 2.6 | 2.8

7. Secondary Outcome: Number of Participants Reported Grade 3+ Adverse Events Within 90 Days After Sublobar Resection
Description: Adverse Events were assessed via the Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0.
Time Frame: 90 days
Population: All Intent-to-Treat (ITT) participants.
Measure: Number; unit: participants
Arm/Group | Arm A (SR) | Arm B (SR + BX)
Number analyzed (Participants) | 114 | 108
participants
  0 - 30 days | 29 | 33
  0 - 90 days | 34 | 40
Statistical Analysis 1: Comparison: Arm A (SR) vs Arm B (SR + BX); Compare the grade 3+ adverse events incidence reported from day 0 to 30 between arms; Test type: Superiority or Other; p = 0.37, Fisher Exact
Statistical Analysis 2: Comparison: Arm A (SR) vs Arm B (SR + BX); Compare the grade 3+ adverse events incidence reported from day 0 to 90 between arms; Test type: Superiority or Other; p = 0.25, Fisher Exact

8. Secondary Outcome: Number of Participants Reported Grade 3+ Respiratory Adverse Events Within 90 Days After Sublobar Resection
Description: The respiratory AE included adult respiratory distress syndrome, aspiration, bronchospasm, bronchostenosis, dyspnea, hypoxia, pleural effusion, pneumonitis, chest tube drainage or leak, prolonged intubation, pulmonary-other, and pneumonia as defined by the CTCAE version 3.0.
Time Frame: 90 days
Population: All Intent-to-Treat (ITT) participants.
Measure: Number; unit: participants
Arm/Group | Arm A (SR) | Arm B (SR + BX)
Number analyzed (Participants) | 114 | 108
participants
  0 - 30 days | 17 | 4
  0 - 90 days | 22 | 6
Statistical Analysis 1: Comparison: Arm A (SR) vs Arm B (SR + BX); Compare the grade 3+ respiratory adverse events incidence reported from day 0 to 30 between arms; Test type: Superiority or Other; p = 0.35, Fisher Exact
Statistical Analysis 2: Comparison: Arm A (SR) vs Arm B (SR + BX); Compare the grade 3+ respiratory adverse events incidence reported from day 0 to 90 between arms; Test type: Superiority or Other; p = 0.31, Fisher Exact

9. Secondary Outcome: Global QOL as Measured Using SF36 at Baseline, Month 3, 12 and 24
Description: Short-form health survey (SF36) consist of 36 items, where scores can be reported as 8 domains of functional health and well-being, or transformed into a physical component summary (PCS) score and a mental component summary (MCS) score. Standardized scores of SF36 PCS and MCS scores were calculated using the mean, SD, and scoring coefficients from the US general population. The standardized scores were then adjusted for age and gender using the mean and SD of the US general population according to age and gender grouping, and employing a linear transformation. Scores <50 indicate below-average health status.
Time Frame: 24 months
Population: Participants who met the eligibility criteria and had SF 36 data at baseline, month 3, 12 or 24.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Arm A (SR) | Arm B (SR + BX)
Number analyzed (Participants) | 108 | 104
units on a scale
  Baseline PCS Scores | 43.2 [21.8 to 62.3] | 41.8 [24.0 to 65.1]
  Baseline MCS Scores | 51.4 [12.2 to 68.6] | 50.5 [17.8 to 69.4]
  Month 3 PCS Scores | 43.2 [19.5 to 61.3] | 42.4 [27.4 to 65.9]
  Month 3 MCS Scores | 51.8 [22.2 to 68.7] | 52.2 [17.6 to 64.0]
  Month 12 PCS Scores | 42.8 [18.8 to 60.0] | 42.8 [27.6 to 64.2]
  Month 12 MCS Scores | 52.5 [22.8 to 69.3] | 51.3 [14.0 to 64.3]
  Month 24 PCS Scores | 44.6 [16.0 to 63.0] | 42.4 [28.2 to 64.9]
  Month 24 MCS Scores | 54.1 [16.5 to 69.1] | 51.2 [28.8 to 65.5]

10. Secondary Outcome: Dyspnea as Measured Using SOBQ at Baseline, Months 3, Months 12 and 24
Description: Dyspnea was evaluated using the University of California, San Diego Shortness of Breath Questionnaire (SOBQ). It consists of 24-item on a scale of 0 to 5 with 0=not at all and 5=maximal or unable to do because of breathlessness. The total scores was calculated by summation of the 24 items scores and transformed into 0-100, with 0= poor quality of life , and 100= excellent quality of life..
Time Frame: 24 months
Population: Participants who met the eligibility criteria and had SOBQ data at baseline, month 3, 12 or 24.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Arm A (SR) | Arm B (SR + BX)
Number analyzed (Participants) | 108 | 104
units on a scale
  Baseline SOBQ Scores | 72.9 [5.8 to 100.0] | 70.0 [5.8 to 98.3]
  Month 3 SOBQ Scores | 75.8 [16.7 to 100.0] | 69.2 [20.8 to 100.0]
  Month 12 SOBQ Scores | 72.5 [13.3 to 100.0] | 72.1 [0.0 to 100.0]
  Month 24 SOBQ Scores | 70.8 [4.2 to 100.0] | 63.8 [5.8 to 95.8]

11. Secondary Outcome: FEV1% Measured at Baseline and Month 3
Description: Pulmonary function tests included percentage predicted forced expiratory volume in 1 second (FEV1%) at baseline and month 3 were compared between arms
Time Frame: 3 months
Population: All participants with complete pulmonary function test data at baseline and month 3.
Measure: Median (Full Range); unit: Percentage of Predicted
Arm/Group | Arm A (SR) | Arm B (SR + BX)
Number analyzed (Participants) | 74 | 74
Percentage of Predicted
  Baseline FEV1% | 49 [22 to 117] | 51 [25 to 110]
  Month 3 FEV1% | 53 [24 to 101] | 53 [24 to 104]
Statistical Analysis 1: Comparison: Arm A (SR); Compare the percentage change from baseline to 3-month value for SR arm; Test type: Superiority or Other; p = 0.03, Wilcoxon Signed Rank
Statistical Analysis 2: Comparison: Arm B (SR + BX); Compare the percentage change from baseline to 3-month value for SR + BX arm; Test type: Superiority or Other; p = 0.18, Wilcoxon Signed Rank

12. Secondary Outcome: DLCO% Measured at Baseline and Month 3
Description: Pulmonary function tests included percentage predicted carbon
  > monoxide diffusing capacity of the lung (DLCO%) at baseline and month 3 were compared between arms.
Time Frame: 3 months
Population: All participants with complete pulmonary function test data at baseline and month 3.
Measure: Median (Full Range); unit: Percentage of Predicted
Arm/Group | Arm A (SR) | Arm B (SR + BX)
Number analyzed (Participants) | 74 | 74
Percentage of Predicted
  Baseline DLCO% | 46 [18 to 97] | 46 [10 to 137]
  Month 3 DLCO% | 48 [14 to 144] | 43 [5 to 96]
Statistical Analysis 1: Comparison: Arm A (SR); Compare the percentage change from baseline to 3-month value for SR arm; Test type: Superiority or Other; p = 0.38, Wilcoxon Signed Rank
Statistical Analysis 2: Comparison: Arm B (SR + BX); Compare the percentage change from baseline to 3-month value for SR + BX arm; Test type: Superiority or Other; p = 0.16, Wilcoxon Signed Rank

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Arm A (SR) | Arm B (SR + BX)
Serious Adverse Events (participants affected / at risk) | 8/114 | 4/108
Other Adverse Events (participants affected / at risk) | 45/114 | 50/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (SR) (N=114) | Arm B (SR + BX) (N=108)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Intraoperative neurological injury - NERVES: Recurrent laryngeal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischemia (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (SR) (N=114) | Arm B (SR + BX) (N=108)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac pain (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 2 (2) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Esophageal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 4 (4)
Pain (General disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 2 (2)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8) | 10 (11)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Intraoperative respiratory injury - Lung (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 6 (6)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prolonged intubation after pulmonary resection (>24 hrs after surgery) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ADH abnormal (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
Leukocyte count decreased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Mini mental status examination abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 3 (3)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 (21) | 27 (27)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 10 (10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 3 (3)
Peripheral ischemia (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 6 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes